CLINICAL TRIAL: NCT00420797
Title: A Double-blind, Randomised, Placebo-controlled Study to Evaluate Topical 10% Phenylephrine Gel in the Management of Ileal Pouch Anal Anastomosis (IPAA)-Related Faecal Incontinence
Brief Title: A Study to Evaluate Topical Phenylephrine Gel in the Management of Faecal Incontinence
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated, new protocol to be developed
Sponsor: S.L.A. Pharma AG (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P/PFI/01
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2007-11

CONDITIONS: Faecal Incontinence
Keywords: Faecal seepage; ileal pouch anal anastomosis (IPAA); quality of life; faecal incontinence; ileo-anal pouch construction; phenylephrine hydrochloride gel; IPAA-related faecal incontinence; placebo
MeSH Terms: conditions — Encopresis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 10% Phenylephrine hydrochloride gel

SUMMARY:
The aim of the study is to test the hypothesis that topical application of phenylephrine improves faecal continence and quality of life in subjects with passive faecal incontinence after ileo-anal pouch construction.

DETAILED DESCRIPTION:
Faecal seepage and even frank incontinence at night can be a problem for approximately 30% of patients who have undergone ileal pouch anal anastomosis (IPAA). Nocturnal seepage may be a problem in patients who do not have gross incontinence, or who may even have no incontinence during the day. Although baseline continence during the day is maintained by involuntary control of the internal anal sphincter, this can be supplemented by voluntary contraction of the external sphincter. While sleeping, this supplementary external sphincter effect is lost and internal anal sphincter tone is reduced, leading to seepage. This is obviously distressing and leads some patients to wear a pad to reduce the soiling that may occur.

The primary objective is to determine the effect of 10% phenylephrine hydrochloride gel, applied three times a day, on the change from baseline to the end of study (8 weeks)in the faecal incontinence score (St Mark's) with passive faecal incontinence after ileo-anal pouch construction, compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Incontinence of solid or liquid stool/mucus following ileo-anal pouch construction, at least once per week over the last month
* At least six months must have elapsed since IPAA surgery or six months since closure of a loop ileostomy created during IPAA surgery, whichever is the later
* Aged 18 years or over
* If female, the subject must not be lactating and must be (a) post-menopausal, (b) surgically sterilised, or (c) have a negative pregnancy test result prior to entry into the study and will use adequate contraception for the duration of the study (sterilization of partner, abstinence, an intra-uterine device (IUD), double barrier method or oral hormonal contraception).
* Written informed consent to participate has been provided

NB: Seepage, leakage, soiling of faecal material is regarded as incontinence.

Exclusion Criteria:

* A history of surgery to the anal sphincter complex
* Active pouchitis (determined by clinical examination and macroscopic inflammation on endoscopy. Patients on maintenance antibiotics need not be excluded but their antibiotic dose should remain the same throughout the study)
* Undergone pelvic radiotherapy at any time
* Cardiac or cardiovascular disease, including ischaemic heart disease, history of stroke, cerebral arteriosclerosis, aneurysm, tachycardia or hypertension
* Hyperthyroidism or diabetes mellitus
* Crohn's disease (indeterminate colitis is not an exclusion criterion)
* The use of α- or β-adrenoceptor agonists (other than inhaled β-adrenoceptor agonists) or antagonists, other sympathomimetics or any cardiovascular drugs during the study (including eyedrops, nasal drops and OTC cold cures containing phenylephrine or pseudoephedrine)
* The use of mono-amine oxidase inhibitors or tricyclic antidepressants in the 4 weeks prior to the first dose of study medication or during the study
* Any mental or other impairment which, in the investigator's opinion, would render them unlikely to be able to comply with the requirements of the study
* Considered by their physician unlikely to be able to comply with the protocol
* Participation in a clinical trial within the past three months
* Known hypersensitivity to phenylephrine or excipients
* History of drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-02; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variable will be the change from baseline to the end of study in the faecal incontinence score (St Mark's)

SECONDARY OUTCOMES:
Efficacy:
Number of daytime faecal incontinence episodes of liquid/mucus and solid stool
Number of nights with nocturnal incontinence episodes of liquid/mucus and solid stool
Number of incontinence episodes of gas
Faecal incontinence quality of life scale
Subject satisfaction with treatment
Subject assessment of overall change from baseline
Loperamide or other constipating agent usage
Anal manometry measurements
Safety:
AEs
Blood pressure
Pulse rate
Changes in other physical examination findings
Changes in biochemical or haematological markers

CONTACTS AND LOCATIONS:
Overall Officials: Susan Clark, MD FRCS, Principal Investigator — St Mark's Hospital, The North West London Hospitals NHS Trust
Locations (1):
- St Mark's Hospital, Harrow, Middlesex, United Kingdom